CLINICAL TRIAL: NCT04129034
Title: Safety and Initial Feasibility of Using the Neurolyser XR Device for the Treatment of Axial Chronic Low Back Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: FUSMobile Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LBP-002
Record Dates: First submitted 2019-10-11; First posted 2019-10-16 (Actual); Last update posted 2022-12-01 (Actual); Status verified 2022-11

CONDITIONS: Facet Syndrome of Lumbar Spine
Keywords: chronic low back pain; zygapophyseal joint syndrome; Facet syndrome

STUDY DESIGN:
Intervention Model Description: Single arm, non-randomized
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): Thermal ablation of the medial nerve branch using High Intensity Focused Ultrasound
  Interventions: Device: Neurolyser XR

INTERVENTIONS:
Device: Neurolyser XR — Non-Invasive Thermal Ablation of the Medial Branch Nerves

SUMMARY:
Single arm pilot study to evaluate the safety and initial feasibility of the Neurolyser XR, a high intensity focused ultrasound device, for non-invasive treatment of axial chronic low back pain

DETAILED DESCRIPTION:
Study design: Prospective, single arm

Timeline: six month enrollment period and 6 months follow-up period.

Sites: The study will be conducted at five sites in Canada: McGill University, Toronto Western, Silver Medical Group, Precision Sport & Spine, Kinetix Integrated Orthopaedic & Regenerative Medicine

Study population: Thirty adult patients diagnosed with facet related low back pain.

Primary study objective: Safety and efficacy of the Neurolyser XR for the treatment of chronic low back pain secondary to zygapophyseal joint syndrome.

Safety is measured by the incidence and severity of treatment related adverse events.

Efficacy is measured by the changes in pain severity at the treatment area, using a numerical rating scale (NRS), of 0 to 10 between baseline and 6 months.

ELIGIBILITY:
Inclusion Criteria:

1. Adult male and females >55 years of age legally able and willing to participate in the study and come for follow-up visits
2. Able and willing to fill the research questionnaires and to communicate with investigator and research team
3. Patient with bilateral or unilateral low back pain of > 6 months duration
4. Patients whose back pain is alleviated by recumbency or comfortable sitting position
5. Patients presenting with a) a positive (>70% pain relief) to a previous, single or double, L1 to L5 lumbar medial branch block (within the last 12 months) and / or b) with a positive (>70% pain relief lasting more than 6 months) to a previous lumbar facet thermal radiofrequency denervation.
6. Average pain score of 6 or higher in the last month, (on 0-10 scale).

Exclusion Criteria:

1. Pregnant or breastfeeding patient
2. Patients younger than 55 or older than 85 years
3. Patients presenting with neurological deficits (including lumbosacral radiculopathy but not solitary radicular pain).
4. Patients with history of lumbosacral spine surgery excluding previous lumbar radiofrequency neurotomy
5. Patients who have had lumbar radiofrequency neurotomy in the past 6 months
6. Patients with the presence of metal hardware or other foreign objects at the lumbosacral spine
7. Patients with history of lumbar spine pathology that may increase procedural risk and / or influence symptoms and / or generate unrelated adverse event, (per the discretion of the study PI)
8. Patients unable to understand and complete the research questionnaires in the official language used within the particular sites' location.
9. Patients presenting with any severe medical condition preventing the patient from safely and effectively being treated in the study or reporting study outcome per PI decision.
10. Patient with extensive scarring of the skin and tissue overlying the treatment area.
11. Patients enrolled in or planned to be enrolled in another clinical trial during the duration of this research project
12. Any patients with an uncontrolled coagulopathy
13. Patients with known osteoporosis with absolute risk of spinal fracture of >10% over 10 years will be excluded
14. Any patients with a history of malignant disease in the past five years
15. Patients with rheumatologic diseases causing spine pain that are currently receiving active treatment including steroids, disease modifying drugs, biological agents or immunosuppressants.
16. Patients known for concomitant psychiatric disorders, excluding mood disorders.
17. Patients presenting with concomitant mood disorders (deemed severe by the research physician).
18. Patients with a first-degree family member already enrolled in this study.
19. Patient who is scheduled for any interventional/surgical procedure within 3 months from screening date
20. Patients diagnosed with co-morbid multifocal chronic pain (e.g., fibromyalgia)

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-09-24 (Actual); Primary Completion 2022-10-26 (Actual); Study Completion 2023-03-26 (Estimated)

PRIMARY OUTCOMES:
NRS | Time Frame: Base line, 2 days 1, 2 & 4 weeks, 3 & 6 months after procedure
  Change in average pain score as measured by a numeric rating scale from 0 (no pain) to 10, worst possible pain
Procedure and Device Safety at six months as measured by measured by the incidence and severity of treatment related adverse events | Time Frame: 6 months after procedure
  Safety will be measured by the incidence and severity of treatment related adverse events

SECONDARY OUTCOMES:
Lesion Size | 2 days post procedure
  Lesion size and location as shown in MRI Image, 2 days post treatment.
Oswestry Disability Index (ODI) | Time Frame: Base line, 1, & 4 weeks, 3 & 6 months after procedure
  Low Back Pain Questionnaire (Range: 0% to 100%)
Short Form 12 (SF-12) | Time Frame: Base line, 1, & 4 weeks, 3 & 6 months after procedure
  A multipurpose short form survey with 12 questions (Range: 0 to 100)
Patient Global Impression of Change (PGIC) | Time Frame: Base line, 1, & 4 weeks, 3 & 6 months after procedure
  Patient Global Impression of Change (Range: 1 to 7)
Procedure and Device Safety as measured by measured by the incidence and severity of treatment related adverse events | Time Frame: Base line, Procedure day, 2 days 1, 2 & 4 weeks, 3 & 6 months after procedure
  Safety will be measured by the incidence and severity of treatment related adverse events

CONTACTS AND LOCATIONS:
Locations (5):
- Canada (5):
  - Kinetix Medicine, Vancouver, British Columbia
  - Precision Sport & Spine, Oakville, Ontario
  - Silver Medical Group, Toronto, Ontario
  - Toronto Western, Toronto, Ontario
  - Alan Edwards Pain Management Unit - Montreal General Hospital, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gofeld M, Smith KJ, Bhatia A, Djuric V, Leblang S, Rebhun N, Aginsky R, Miller E, Skoglind B, Hananel A. Fluoroscopy-guided high-intensity focused ultrasound neurotomy of the lumbar zygapophyseal joints: a prospective, open-label study. Reg Anesth Pain Med. 2025 Jun 10;50(6):464-470. doi: 10.1136/rapm-2024-105345. PMID 38580339